CLINICAL TRIAL: NCT06369948
Title: Quality Of Recovery After Pericapsular Nerve Group (PENG) Block For Hip Hemiarthroplasty Under Spinal Anesthesia: A Prospective, Double-Blinded, Randomized Controlled Trial
Brief Title: Quality Of Recovery After Pericapsular Nerve Group (PENG) Block For Hip Hemiarthroplasty Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Atef Mohamed mahmoud, Associate professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M703
Record Dates: First submitted 2024-03-31; First posted 2024-04-17 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hip Hemiarthroplasty
Keywords: PENG block; pain management; spinal Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion; Bupivacaine; Injections

STUDY DESIGN:
Intervention Model Description: We will include 60 patients who will undergoe elective hip hemiarthroplasty. Patients will be divided into two groups randomized by computer generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the block.
  Pericapsular Nerve Group (PENG) Block (P group) includes 30 patients who will receive a PENG block.
  Control group (C group) includes 30 patients who will not receive a PENG block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be divided into two groups randomized by computer generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the block.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pericapsular Nerve Group (PENG) Block (P group) (Experimental): Patients who will undergo elective hip hemiarthroplasty and receive the Pericapsular Nerve Group (PENG) block postoperatively.
  Interventions: Procedure: Pericapsular Nerve Group (PENG) Block; Drug: bupivacaine 0.5% injection
- Control group (C group) (Active Comparator): Patients who will undergo elective hip hemiarthroplasty without receiving a PENG block.
  Interventions: Procedure: elective hip hemiarthroplasty without receiving a PENG block.

INTERVENTIONS:
Procedure: Pericapsular Nerve Group (PENG) Block — The PENG block will be performed with the patient in the supine position. A linear high-frequency ultrasound probe (GE LOGIQ/P7 ultrasound, korea/ L6-12RS probe) is initially placed in a transverse plane over the anterior inferior iliac spine (AIIS); the probe is turned slightly medial until the hyperechoic continuous shadow of the iliopubic eminence (IPE). The target will be the plane between the psoas tendon and pubic ramus. The skin puncture site will be anesthetized using lidocaine 2% after skin disinfection and draping. A 22-gauge, 100 mm echogenic needle (Spinocan, B. Braun Melsungen AG, Germany) will be inserted in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, 25 mL of the local anesthetic solution (bupivacaine 0.5%) was injected in 5 mL increments while observing for adequate fluid spread in this plane.
  Arms: Pericapsular Nerve Group (PENG) Block (P group)
Procedure: elective hip hemiarthroplasty without receiving a PENG block. — elective hip hemiarthroplasty without receiving a PENG block.
  Arms: Control group (C group)
Drug: bupivacaine 0.5% injection — bupivacaine 0.5% injection
  Arms: Pericapsular Nerve Group (PENG) Block (P group)

SUMMARY:
Patients undergoing hip hemiarthroplasty can benefit significantly from regional anesthesia in terms of pain management and recovery . There is a wide range of regional anesthetic techniques. The most common in this anatomical region and those with the greatest published research are fascia iliac block, lumbar plexus block, and femoral nerve block . Alternative methods include lateral femoral cutaneous nerve and selective obturator nerve infiltration blocks. Novel techniques, including local infiltration analgesia and quadratus lumborum block, have been reported.

While femoral nerve and lumbar plexus blocks are two common opioid-sparing regional anesthetic procedures that are successful, they come with a risk of undesired lower limb muscle weakness . On the other hand, the fascia iliac block does not always offer sufficient pain relief following hip surgery. The important landmarks targeted on the hip joint branches from the femoral nerve and the auxiliary obturator nerve may now be identified thanks to a recent anatomical study on hip innervation .

This led to the discovery of a novel localized anesthetic treatment termed pericapsular nerve group block (PENG), which blocks these nerves to target the hip's anterior capsule. The PENG block has been suggested as a successful motor-sparing block for hip hemiarthroplasty . The objective of the current study is to evaluate the efficacy of the pericapsular nerve group block (PENG) for the reduction of opioid consumption and management of postoperative pain after hip hemiarthroplasty.

DETAILED DESCRIPTION:
This study will be performed in the Fayoumi University Hospital after approval by the local Institutional Ethics Committee and local institutional review board. The study design will be a double-blinded, randomized controlled study trial. The researcher will inform the participants about the objectives of the study, the examination, and the investigation that will be done. Also, the confidentiality of their information and their right not to participate in the study. Written informed consent will be obtained from all patients included in the study.

The study will include 60 patients who will undergo elective hip hemiarthroplasty. Patients will be divided into two groups randomized by computer generated random numbers that will be placed in separate opaque envelopes that will be opened by study investigators just before the block.

Pericapsular Nerve Group (PENG) Block (P group) includes 30 patients who will receive a PENG block.

Control group (C group) includes 30 patients who will not receive a PENG block. A full medical history will be taken from the included patients, including demographic data (age, body mass index , weight, gender), general medical history (Diabetes, Hypertension, medication use), anesthesia, and previous surgeries. The patients' fasting durations will be 8 hours for solids and 2 hours for clear liquids. All patients will be assessed Preoperative for VAS score. All patients were monitored by 5 lead ECG, pulse oximetry, non-invasive blood pressure and an intravenous access will be established.

The technique of spinal anesthesia will be standardized for all patients, an attending anesthesiologist will use a 25-gauge Quincke spinal needle (Spinocan, B. Braun Melsungen AG, Germany) to induce spinal anesthesia in the L3/4 or L4/5 vertebral interspace. Throughout the course of the trial, the attending anesthesiologist will chose the dosages of 0.5% hyperbaric bupivacaine (10 to 15 mg) and fentanyl (15 mcg), aiming for a sensory block at the T4 level. The patient will be placed in the sitting or left lateral position while the spinal injection is given over a period of 15 to 30 seconds. Three minutes following the spinal injection, the sensory block was evaluated with a cold and pinprick test. The patient will be placed in a supine position, neutral-head resting posture in the operating area as standard monitors that mentioned before .

Data will be gathered, coded to make data manipulation easier, double-entered into Microsoft Access, and will be analyzed using SPSS software version 22 running on Windows 7 (SPSS Inc., Chicago, IL, USA). Simple descriptive analysis will use percentages and numbers for qualitative data, arithmetic means for measuring central tendency, and standard deviations for quantifying dispersion for parametric quantitative data.

- For quantitative data: Independent samples t-test will be used to compare quantitative measures between two independent groups Paired t-test will be used to compare two dependent quantitative data.

* For qualitative data The Chi-square test will be used to compare two of more than two qualitative groups.
* Sensitivity and specificity test for testing a new test with ROC curve "Receiver Operating Characteristic".

  * The P-value< 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* - patients 18 years old or older with ASA physical status 1-3, patients who had no contraindications for spinal anesthesia, and patients undergoing elective surgery.

Exclusion Criteria:

* Patients with ASA physical status 4 or above.
* Pre-existing anatomical or neurological deﬁcits in the lower extremity.
* Intolerance or allergy to local anesthetics.
* Narcotic dependency.
* Coagulopathy or using antiplatelet or anticoagulant medications.
* Neuromuscular diseases.
* Psychiatric illnesses (schizophrenia, bipolar, uncontrolled anxiety or depression).
* Systemic infections or infections at site of injection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption post operative | from zero hour and at time intervals: 30 minutes, 1hour, 3 hour, 6 our., 12 hour, 24 hour, 48 hour, and 36 hour after block administration
  total dose of any opioid drug used for pain control postoperative

SECONDARY OUTCOMES:
2) a Visual Analogue Scale (VAS) ranging from zero (no pain) to 10 (severe pain) for dynamic and static pain | at time intervals: 30 minutes, 1hour, 3 hour, 6 hour, 12 hour, 24 hour, 48 hour, and 72 hour. after block administration
  Degree of pain as measured by fascial expression with rang from 0 for no pain to 10 for sever pain
3) Time to first opioid use | first 24 hour after block administration
  time taken till first dose of opioid drugs to control pain after 24 hour of block administration
4) Ability to perform physiotherapy | 1 year
  time taken until the participant able to perform physiotherapy in first 24 hour after block administration
5) Opioid-related side effects. | 1 year
  side effects of opioids used for pain control after surgery
6) Total length stay of hospital | 1 year
  time of stay of the participant in the hospital after surgery and block administration
7) Complications of local anesthetic toxicity | 1 year
  complication of local anesthetic drug injected in the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Atef Mohamed Sayed, MS.C, Principal Investigator — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University Hospital, El Fayoum Qesm, Fayoum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meng Y, Deng B, Liang X, Li J, Li L, Ou J, Yu S, Tan X, Chen Y, Zhang M. Effectiveness of self-efficacy-enhancing interventions on rehabilitation following total hip replacement: a randomized controlled trial with six-month follow-up. J Orthop Surg Res. 2022 Apr 10;17(1):225. doi: 10.1186/s13018-022-03116-2. PMID 35399102
- [Background] van Drongelen S, Kaldowski H, Tarhan T, Assi A, Meurer A, Stief F. Are changes in radiological leg alignment and femoral parameters after total hip replacement responsible for joint loading during gait? BMC Musculoskelet Disord. 2019 Nov 10;20(1):526. doi: 10.1186/s12891-019-2832-5. PMID 31707985
- [Background] Zaballa E, Dennison E, Walker-Bone K. Function and employment after total hip replacement in older adults: A narrative review. Maturitas. 2023 Jan;167:8-16. doi: 10.1016/j.maturitas.2022.09.005. Epub 2022 Sep 14. PMID 36302339
- [Background] Chen L, Chen G. The Effect of Resistance Training on the Function after Hip Replacement: A Meta-analysis of Randomized Controlled Trials. Z Orthop Unfall. 2021 Aug;159(4):383-390. doi: 10.1055/a-1154-8949. Epub 2020 Dec 9. PMID 33296947
- [Background] Domingue G, Warren D, Koval KJ, Riehl JT. Complications of Hip Hemiarthroplasty. Orthopedics. 2023 Jul-Aug;46(4):e199-e209. doi: 10.3928/01477447-20230125-06. Epub 2023 Jan 30. PMID 36719411
- [Background] Tsai MC, Ng YY, Chen WM, Tsai SW, Wu SC. The effects of cement fixation on survival in elderly patients with hip hemiarthroplasty: a nationwide cohort study. BMC Musculoskelet Disord. 2019 Dec 27;20(1):628. doi: 10.1186/s12891-019-3013-2. PMID 31881878
- [Background] Lee C, Freeman R, Edmondson M, Rogers BA. The efficacy of tranexamic acid in hip hemiarthroplasty surgery: an observational cohort study. Injury. 2015 Oct;46(10):1978-82. doi: 10.1016/j.injury.2015.06.039. Epub 2015 Jul 6. PMID 26190627
- [Background] Pala E, Trono M, Bitonti A, Lucidi G. Hip hemiarthroplasty for femur neck fractures: minimally invasive direct anterior approach versus postero-lateral approach. Eur J Orthop Surg Traumatol. 2016 May;26(4):423-7. doi: 10.1007/s00590-016-1767-x. Epub 2016 Mar 30. PMID 27026091
- [Background] Spaans EA, Koenraadt KLM, Wagenmakers R, Elmans LHGJ, van den Hout JAAM, Eygendaal D, Bolder SBT. Does surgeon volume influence the outcome after hip hemiarthroplasty for displaced femoral neck fractures; early outcome, complications, and survival of 752 cases. Arch Orthop Trauma Surg. 2019 Feb;139(2):255-261. doi: 10.1007/s00402-018-3076-9. Epub 2018 Nov 27. PMID 30483916
- [Background] Moore BF, Lachiewicz PF. Corrosion and adverse tissue reaction after modular unipolar hip hemiarthroplasty. Arthroplast Today. 2017 Feb 21;3(4):207-210. doi: 10.1016/j.artd.2017.01.002. eCollection 2017 Dec. PMID 29204481
- [Background] Verzellotti S, Candrian C, Molina M, Filardo G, Alberio R, Grassi FA. Direct anterior versus posterolateral approach for bipolar hip hemiarthroplasty in femoral neck fractures: a prospective randomised study. Hip Int. 2020 Nov;30(6):810-817. doi: 10.1177/1120700019872117. Epub 2019 Aug 26. PMID 31450987
- [Background] Short AJ, Barnett JJG, Gofeld M, Baig E, Lam K, Agur AMR, Peng PWH. Anatomic Study of Innervation of the Anterior Hip Capsule: Implication for Image-Guided Intervention. Reg Anesth Pain Med. 2018 Feb;43(2):186-192. doi: 10.1097/AAP.0000000000000701. PMID 29140962
- [Background] Morrison C, Brown B, Lin DY, Jaarsma R, Kroon H. Analgesia and anesthesia using the pericapsular nerve group block in hip surgery and hip fracture: a scoping review. Reg Anesth Pain Med. 2021 Feb;46(2):169-175. doi: 10.1136/rapm-2020-101826. Epub 2020 Oct 27. PMID 33109730
- [Background] Kupeli I, Yazici Kara M. Anesthesia or analgesia? New block for shoulder surgery: pericapsular nerve group block. Braz J Anesthesiol. 2022 Sep-Oct;72(5):669-672. doi: 10.1016/j.bjane.2021.05.009. Epub 2021 Jun 9. PMID 34118263
- [Background] Gullupinar B, Saglam C, Unluer EE, Ayvat P, Ozturk K, Gul M, Tandon S. Effectiveness of pericapsular nerve group block with ultrasonography in patients diagnosed with hip fracture in the emergency department. Ulus Travma Acil Cerrahi Derg. 2022 Jun;28(6):832-838. doi: 10.14744/tjtes.2022.67817. PMID 35652877
- [Background] Farag A, Hendi NI, Diab RA. Does pericapsular nerve group block have limited analgesia at the initial post-operative period? Systematic review and meta-analysis. J Anesth. 2023 Feb;37(1):138-153. doi: 10.1007/s00540-022-03129-5. Epub 2022 Nov 7. PMID 36342537
- [Background] Wang Y, Wen H, Wang M, Lu M. The Efficiency of Ultrasound-Guided Pericapsular Nerve Group Block for Pain Management after Hip Surgery: A Meta-analysis. Pain Ther. 2023 Feb;12(1):81-92. doi: 10.1007/s40122-022-00463-0. Epub 2022 Dec 8. PMID 36481969
- [Background] Mysore K, Sancheti SA, Howells SR, Ballah EE, Sutton JL, Uppal V. Postoperative analgesia with pericapsular nerve group (PENG) block for primary total hip arthroplasty: a retrospective study. Can J Anaesth. 2020 Nov;67(11):1673-1674. doi: 10.1007/s12630-020-01751-z. Epub 2020 Jul 13. No abstract available. PMID 32661723
- [Background] Ueshima H, Otake H. RETRACTED: Clinical experiences of pericapsular nerve group (PENG) block for hip surgery. J Clin Anesth. 2018 Dec;51:60-61. doi: 10.1016/j.jclinane.2018.08.003. Epub 2018 Aug 8. No abstract available. PMID 30096522 (Retraction: PMID 35393178 J Clin Anesth. 2022 Aug;79:110722)
- [Background] Kukreja P, Uppal V, Kofskey AM, Feinstein J, Northern T, Davis C, Morgan CJ, Kalagara H. Quality of recovery after pericapsular nerve group (PENG) block for primary total hip arthroplasty under spinal anaesthesia: a randomised controlled observer-blinded trial. Br J Anaesth. 2023 Jun;130(6):773-779. doi: 10.1016/j.bja.2023.02.017. Epub 2023 Mar 22. PMID 36964012